CLINICAL TRIAL: NCT03330080
Title: Examining Sleep and Family Functioning in Pediatric Craniopharyngioma Using Ecological Momentary Assessment
Brief Title: Examination of Sleep and Family Functioning in Pediatric Craniopharyngioma Patients
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: SAFF
Record Dates: First submitted 2017-10-31; First posted 2017-11-06 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Craniopharyngioma
Keywords: Ecological momentary assessment; Sleepiness; Fatigue; Endocrinopathy; Family functioning
MeSH Terms: conditions — Craniopharyngioma; Sleepiness; Fatigue; Endocrine System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ecological momentary assessment (EMA): The ecological momentary assessment (EMA) will be used for participants to complete surveys from home on two occasions each day over seven days.

SUMMARY:
Pediatric craniopharyngioma patients experience significant endocrine and sleep dysregulation difficulties. Sleep is a crucial part of children's healthy development, and sleep difficulties are associated with severe functional morbidity. Insufficient sleep, excessive daytime sleepiness, and poor sleep quality have all been significantly related to academic, behavioral, and emotional functioning in children and adolescents. Ecological momentary assessments (EMA) will be used to collect observational data.

EMA data will be collected twice daily for one week. For the morning EMA administration, participants will be asked about their sleep. During the evening administration, participants will be asked about their daytime sleepiness, overall well-being, and family functioning. Covariates also administered during the evening administration include medication administration (Y/N) and total screen time. At the end of the EMA data collection period (on day 7 OR 8), participants will be sent a survey asking them to report - anonymously - their overall experience and satisfaction with the EMA data collection method.

DETAILED DESCRIPTION:
After recruitment and informed consent/assent is obtained for the current study, participants will be asked to complete a questionnaire battery online (via REDCap) assessing sleep habits, daytime sleepiness, family routines, family functioning, and overall quality of life in the past six months. The relationship between subjective sleep ratings obtained from the parent craniopharyngioma study at St. Jude (RT2CR) at diagnosis and 3 months later (T1 and T2) and family functioning/routines at the follow-up study (T3) will be assessed. The researchers have permission to use data for all participants who consent to participate in this follow-up EMA study.

Children will be sent electronic surveys two times per day (i.e., morning and evening) for seven days using Ilumivu software (https://ilumivu.com/mema-demo). Ilumivu is an established EMA tool that offers an in-mobile app for participants to respond to questionnaires in real time with limited burden. This application will send notifications to participants to remind them to complete surveys and record response times for each survey.

ELIGIBILITY:
Inclusion Criteria:

* Craniopharyngioma diagnosis
* Access to smartphone or a tablet
* Agreement to download Ilumivu application
* The ability for the participant to answer questionnaires (i.e., no cognitive or developmental diagnoses that would preclude understanding and completing child self-report questionnaires)
* Age between 8 and 18 years old at the time of enrollment onto St. Jude protocol RT2CR.
* Participated in sleep study component of RT2CR

Exclusion Criteria:

* Limited English proficiency as evidenced by an inability to read and respond to EMA survey questions
* Visual or sensorimotor impairment (e.g., loss of sight)

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants for the proposed study will be children who participated in the parent study (ages 8-18 at the time of enrollment on RT2CR) and have an ongoing relationship with the study team. They will be contacted during their follow-up clinic visits and invited to participate in this additional study. Parental consent and participant assent (if age <18) or consent (if age ≥18) for the proposed study will be obtained in-person.
  Two institutions will collaborate in the proposed project: St. Jude Children's Research Hospital (SJCRH) and Virginia Commonwealth University (VCU), however, recruitment, patient enrollment, and data collection will only take place at St. Jude.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2019-01-29 (Actual); Study Completion 2019-01-29 (Actual)

PRIMARY OUTCOMES:
Rate of participation | Once at enrollment
  Study feasibility will be assessed by calculating the participation rate as follows: the number of participants who agree to participants divided by the number who are approached to participate.

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Crabtree, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St . Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: clinical Trials Open at St. Jude — http://www.stjude.org/protocols